CLINICAL TRIAL: NCT05362045
Title: Bioequivalence Study of a Single Dose of 15-mg Mavacamten Capsule Versus a Single Dose of 3 x 5-mg Mavacamten Capsules in Healthy Participants
Brief Title: A Study to Evaluate the Effects on the Single-Dose Drug Levels of Mavacamten in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV027-070
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Healthy Participants
Keywords: Mavacamten; Healthy Participants; Bioequivalence; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mavacamten- Dose A (Experimental)
  Interventions: Drug: Mavacamten
- Mavacamten- Dose B (Experimental)
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — Specified dose on specified days
  Other Names: BMS-986427; MYK-461

SUMMARY:
The purpose of this study is to evaluate the effects on the single-dose drug levels of mavacamten in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 32 kg/m^2, inclusive, at the Screening Visit
* Healthy, as determined by physical examination, vital signs, electrocardiograms (ECGs), and clinical laboratory assessments within the normal range at the screening visit and/or on Day -1

Exclusion Criteria:

* Current or recent (within 3 months of study intervention administration) gastrointestinal disease
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity)

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to approximately 1 month
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration ((AUC(0-T)) | Up to approximately 1 month
Area under the plasma concentration-time curve from time zero extrapolated to infinite time ((AUC(INF)) | Up to approximately 1 month

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to approximately 1 month
Terminal half-life (T-HALF) | Up to approximately 1 month
Number of participants with adverse events (AEs) | Up to approximately 1 month
Number of participants with serious adverse events (SAEs) | Up to approximately 1 month
Number of participants with vital sign abnormalities exceeding predefined thresholds | Up to approximately 1 month
Number of participants with electrocardiogram (ECG) abnormalities | Up to approximately 1 month
Number of participants with physical exam abnormalities | Up to approximately 1 month
Number of participants with clinical laboratory evaluation abnormalities | Up to approximately 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Clinical pharmacology of Miami, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - QPS Springfield, Springfield, Missouri
  - Ppd Phase I Clinic, Austin, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm